CLINICAL TRIAL: NCT04400825
Title: Comparing Dry Needling and Stretching for the Management of Muscle Extensibility in Patients With Hip Osteoarthritis: A Randomized Clinical Trial
Brief Title: Dry Needling Versus Stretching for Muscle Extensibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Luis Ceballos Laita, Ph.D, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIm1955
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis, Hip
Keywords: physiotherapy; stretching; dry needling
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Dry needling of 3 active MTrPs at most.
  Interventions: Other: Dry needling
- Stretching (Active Comparator): Stretching of the main hip flexors (rectus femoris, iliopsoas and tensor fasciae latae)
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — Dry needling of the active MTrPs following the technique described by Hong et al (1994,1995)

SUMMARY:
Hip osteoarthritis (OA) is one of the most prevalent chronic disease in the world. Currently several authors have shown the presence of active myofascial trigger points (MTrP) in the muscles surrounding the hip joint that reproduce the symptoms of the patients with hip OA.

Despite of the beneficial effects that have shown may conservative non-pharmacological treatments, there is a lack of studies evaluating the effects of the conservative treatments on muscle extensibility.

According to the new paradigm about the presence of MTrPs, the investigators decided to conduct a randomized clinical trial to compare the effects of DN intervention and stretching protocol on muscle extensibility in patients with hip OA.

ELIGIBILITY:
Inclusion Criteria:

* unilateral hip OA diagnosed medically with a X-Ray tess and following the American College of Rheumatology Criteria

Exclusion Criteria:

* Secondary osteoarthritis by a traumatism, Paget disease, inflammatory or metabolic disease, congenital diseases etc.
* Vascular or neurological disease.
* Musculoskeletal pathologies in lumbar spine, pelvis or lower limbs
* DN contraindications or fear of needles

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-19 (Actual); Study Completion 2020-07-19 (Actual)

PRIMARY OUTCOMES:
muscle extensibility | Baseline
  the examiners assess the muscle extensibility using an inclinomenter
muscle extensibility | up to 3 weeks
  the examiners assess the muscle extensibility using an inclinomenter

SECONDARY OUTCOMES:
Stiffness | Baseline
  the examiners assess the stiffness using the WOMAC stiffness subscale
Stiffness | up to 3 weeks
  the examiners assess the stiffness using the WOMAC stiffness subscale

CONTACTS AND LOCATIONS:
Locations (1):
- Luis Ceballos Laita, Soria, Spain

IPD SHARING:
Plan to Share IPD: No